CLINICAL TRIAL: NCT03531749
Title: Antioxidant Activity and Lipid Peroxidation Status in Patients HIV+ Supplemented With Microencapsulated of Red Pomegranate
Brief Title: Antioxidant in Patients HIV+ Supplemented With Microencapsulated of Red Pomegranate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma del Estado de Hidalgo (Other)
Collaborators: National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Gabriel Betanzos Cabrera, Professor-Researcher, Universidad Autónoma del Estado de Hidalgo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FSSA2016051
Record Dates: First submitted 2017-11-01; First posted 2018-05-22 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Intervention Model Description: A prospective double-blind randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: A prospective double-blind, randomized clinical trial of microencapsulated of red pomegranate to treat HIV-infected patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HIV+ MRPJ (Experimental): Supplementation with microencapsulated (1g/d) for 90 days
  Interventions: Dietary Supplement: HIV+ MRPJ
- HIV+ ascorbic acid (Experimental): Supplementation with ascorbic acid (1g/d) for 90 days
  Interventions: Dietary Supplement: HIV+ ascorbic acid
- HIV- MRPJ (Experimental): Supplementation with microencapsulated (1g/d) for 90 days
  Interventions: Dietary Supplement: HIV+ MRPJ
- HIV- ascorbic acid (Experimental): Supplementation with ascorbic acid (1g/d) for 90
  Interventions: Dietary Supplement: HIV+ ascorbic acid
- HIV- Control (No Intervention): Unsupplemented
- HIV+ Control (No Intervention): Unsupplemented

INTERVENTIONS:
Dietary Supplement: HIV+ MRPJ — supplemented with (1g/d) MRPJ
  Arms: HIV+ MRPJ; HIV- MRPJ
Dietary Supplement: HIV+ ascorbic acid — Supplemented with (1g/d) AA
  Arms: HIV+ ascorbic acid; HIV- ascorbic acid

SUMMARY:
Human immunodeficiency virus (HIV) infection continues to be a pandemic, Mexico has around 184,000 people infected by this virus. A common metabolic problem for these patients is oxidative stress (OS), which has been related with the progression of the disease and the presence of comorbidities. Pomegranate is a fruit rich in antioxidants, which potentially can inhibit or reduce deleterious metabolic compounds resulting from OS; however; it has never been tested in patients infected with HIV. The present project was done in patients HIV+ from state of Hidalgo in order to see the effects of microencapsulated red pomegranate juice (MRPJ) and ascorbic acid (AA) on antioxidant activity and lipid peroxidation both biomarkers of oxidative stress. Sixty subjects were recruited, 30 HIV positive (HIV+) and 30 HIV negative (HIV-). Three subgroups (n=10) were formed from each group: 1) supplemented with (1g/d) MRPJ; 2) supplemented with 1g/d AA; and 3) control group (unsupplemented). The intervention lasted 90 days and blood samples were taken four times: at the beginning and every 30 days. Antioxidant activity in the blood serum was measured by the DPPH (2,2-diphenyl-1-picrylhydrazyl) and ABTS + (2,2'-azino-bis(3-ethylbenzothiazoline-6-sulphonic acid) methods while lipid peroxidation by malondialdehyde (MDA) levels which was measured by TBARS method. The baseline results showed a significant decrease of antioxidant activity in HIV+ groups compared to the HIV- groups, although there was no significant difference in lipid peroxidation, as measured by MDA assay levels. Several studies suggest that the reduction of antioxidant activity is a consequence of the infection and the antiretroviral treatment, although the organism tries to reestablish it unbalance it usually fails, thus (OS) is significant in these patients. The groups that received AA had antioxidant activity greater than the MRPJ treated. MRPJ treatment, however, the groups that received MRPJ had significantly reduced lipid peroxidation. Reduced lipid peroxidation could have more beneficial effects on HIV+ subjects since the reduction of markers of OS, such as lipid peroxidation, has been associated with reductions in the risk of death from HIV.

DETAILED DESCRIPTION:
Since Patients HIV+ suffer oxidative stress, microencapsulated of red pomegranate juice will be evaluated for decreasing oxidative stress in HIV+ patients it will be compared with patients treated with ascorbic acid. The supplementation will take 90 days and blood samples were taken four times: at the beginning of the study and every 30 days thereafter. Antioxidant activity in the blood serum was measured by the DPPH and ABTS+ methods lipid peroxidation was measured as stress oxidative markers

ELIGIBILITY:
Inclusion criteria:

* Over 18 years
* Having a positive HIV diagnosis
* Having antiretroviral treatment
* Status of one of the following clinical categories A1, A2, B1 and B2 at the time of the study start,
* Residents of the city of Pachuca

Exclusion Criteria:

* Subjects taking antioxidants
* Pregnant women.
* Subjects taking of angiotensin-converting enzyme inhibitors (e.g.captopril or enalapril).
* subjects who do not comply with at least 95% of the adherence of the supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-01; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Biochemical analyses to determine antioxidant capacity | At 0 time (baseline)
  Four different tests for antioxidant activity were utilized. Plasma antioxidant capacity, catalase, H2O2, and TBARS

SECONDARY OUTCOMES:
Biochemical analyses to determine antioxidant capacity | 30 days after intervention
  Four different tests for antioxidant activity were utilized. Plasma antioxidant capacity, catalase, H2O2, and TBARS

IPD SHARING:
Plan to Share IPD: No